CLINICAL TRIAL: NCT01633957
Title: Academic Leader，Head of Cardiac Surgery,Principal Investigator, Clinical Professor
Brief Title: A Trial of Genotype-based Warfarin Initiation in Patients With Mechanical Prosthetic Heart Valve
Acronym: SYSU-WARFA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xi Zhang (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor-Investigator, Xi Zhang, Head of cardiac surgery, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYSU-XZ001
Record Dates: First submitted 2012-06-20; First posted 2012-07-06 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Anticoagulation Treatment Overdose; Heart Valve Diseases
Keywords: anticoagulation; bleeding; CYP2C9; CYP4F2; VKORC1; warfarin dosing; Heart Valve Diseases; pharmacogenomics
MeSH Terms: conditions — Heart Valve Diseases; Hemorrhage; Vitamin K-Dependent Clotting Factors, Combined Deficiency Of, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Genotype-based Warfarin Initiation (Experimental)
  Interventions: Other: Genotype-based Warfarin Initiation model
- clinical factor-based warfarin initiation (Active Comparator)
  Interventions: Other: clinical factor-based warfarin initiation model

INTERVENTIONS:
Other: Genotype-based Warfarin Initiation model — Based on previous retrospective study,investigators established a genotype-based warfarin model to estimate the drug dosage.
  Arms: Genotype-based Warfarin Initiation
Other: clinical factor-based warfarin initiation model — Based on previous retrospective study,investigators established a clinical factor-based warfarin model to estimate the drug dosage.
  Arms: clinical factor-based warfarin initiation

SUMMARY:
Until very recently, warfarin is still the best drug of choice for long-term anticoagulation for patients with mechanical prosthetic heart valve. However, the complication of warfarin account for 75 percent of the whole complication after the mechanical prosthetic heart valve replacement.

Interindividual variation in warfarin dose is mediated by multiple factors.Advanced models using combinations of clinical attributes and genetic factors(CYP2C9, VKORC1, and CYP4F2) explain 50-75% of variability in warfarin dose requirements.These warfarin dosing models have the potential to improve patient safety by reducing or eliminating serious adverse events. The investigators conducted a prospective, randomized, blinded, two arm trial to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* the first time to receive elective mitral and/or aortic mechanical prosthetic valve replacement
* willing to join in the clinical trial and comply with the protocol.

Exclusion Criteria:

* other ethnic groups than Han
* previously receive any other cardiac surgery
* emergent surgery
* simultaneously carry out other cardiac surgeries,such as CABG
* age younger than 18y or older than 65 year
* drug abuser and wine abuser
* any malignancy
* moderate or severe hepatic or kidney insufficiency
* any thyroid disease
* the history of warfarin or VitK consumption 2 week before the surgery
* any hematological disease or history of bleeding
* combination with any drugs that significantly influence warfarin other than Cordarone
* pregnancy
* any contraindication of warfarin
* infectious endocarditis
* advanced valvular disease
* pathological obesity
* psychological disease
* any patient having joined in other clinical trial in the previous 30d
* basic INR > 1.4

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
time to steady dosage | from seven days after the operation to thirty days after the operation
Time in Therapeutic Range | from five days after the operation to thirty days after the operation

SECONDARY OUTCOMES:
first time to treatment window | from five days after the operation to thirty days after the operation
the ratio of INR≥3.0 and INR≤1.5 | from five days after the operation to thirty days after the operation
the monitoring frequency of INR | 30 days after the operation
the whole-cause mortality | 30 days after the operation
major bleeding event | 30 days after the operation
major thrombosis rate | 30 days after the operation
absolute difference between the stable dose and initial dose | 30 days after the operation
the frequency of dosage change | 30 days after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Xi Zhang, MD., Study Director — First Affiliated Hospital, Sun Yat-Sen University; Zhe Xu, MD.,PHD., Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The first affiliated hospital of Sun Yat Sen University, Guangzhou, Guangdong, China

REFERENCES:
- See also: one of the best warfarin dose model — http://warfarindosing.org/Source/Home.aspx